CLINICAL TRIAL: NCT00643903
Title: The Balance Project - RCT of an HIV Treatment Side Effects Coping Intervention
Brief Title: Effectiveness of Coping Training for People With HIV Experiencing Treatment Side Effects (The Balance Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01MH068208 (NIH); R01MH068208 (NIH); DAHBR 9A-ASGA
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: Side Effects; Adherence; Coping; HIV; AIDS; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive five individual sessions of coping effectiveness training.
  Interventions: Behavioral: Cognitive behavioral coping effectiveness training
- 2 (Active Comparator): Participants will receive standard care and one delayed group workshop of coping effectiveness training.
  Interventions: Behavioral: Standard care; Behavioral: Single group workshop on coping effectiveness training

INTERVENTIONS:
Behavioral: Cognitive behavioral coping effectiveness training — Coping effectiveness training will include five individual 90-minute counseling sessions. The sessions will focus on coping with stress, dealing with medication side effects, and staying on track with medications.
  Arms: 1
Behavioral: Standard care — Participants will receive standard of care for HIV infections.
  Arms: 2
Behavioral: Single group workshop on coping effectiveness training — Participants will attend one group workshop covering the same material as in the individual sessions. The workshop will be delivered after completion of the Month 18 final assessment.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of cognitive behavioral coping training in improving side effect management and treatment adherence in HIV-infected patients who are taking antiretroviral medications.

DETAILED DESCRIPTION:
HIV is a virus that is transmitted through the exchange of bodily fluids, primarily through sexual intercourse. HIV infections can lead to acquired immunodeficiency syndrome (AIDS), a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. Antiretroviral therapy (ART) has proven to effectively inhibit the replication of HIV and has resulted in a reduction in HIV-related deaths. People infected with HIV who are receiving ART, however, may be confronted with negative physical and emotional side effects. These side effects can impact quality of life (QOL), adherence to medical care, and decisions about health care. Stress and Coping Theory (SCT) is a person-centered approach that considers stressful experiences as person-environment transactions. A cognitive behavioral treatment based upon SCT may help to eliminate or reduce the negative impact of side effects, improve QOL, and maximize benefit from treatment among people living with HIV. This study will evaluate the effectiveness of cognitive behavioral coping training in improving side effect management and treatment adherence in HIV-infected people who are taking ART medications.

This study will involve two phases. Phase 1 will be conducted over 12 months and will include two 1-hour interviews with questions about personal life, family, friends, medications, and medication side effects. After the first interview, participants may be invited to participate in Phase 2, which will last 18 months.

During Phase 2, participants will complete five 2- to 3-hour interviews occurring at baseline and Months 3, 6, 12, and 18. Interviews will include questions about personal life, friends, family, health-related activities, drug-using behaviors, emotions, mental state, and educational background. Participants will be assigned randomly to one of two treatment groups:

* Group 1 participants will receive five individual sessions of cognitive behavioral coping training, beginning after the Month 3 interview. The 90-minute sessions will focus on coping with stress, dealing with medication side effects, and staying on track with medications.
* Group 2 participants will receive standard care and one group session of coping training, which will be held after the Month 18 interview. The group session will cover the same material that is covered in the individual sessions.

After the last follow-up interview, some participants may also be asked to complete an exit interview about thoughts and feelings on study participation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of HIV infection
* Currently receiving ART
* Experiencing ART side effects

Exclusion Criteria:

* Currently enrolled in another trial
* Evidence of psychosis or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-04; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Quality of life | Measured at Month 18

SECONDARY OUTCOMES:
Medication adherence | Measured at Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Mallory O. Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States